CLINICAL TRIAL: NCT04107623
Title: Quantitative Fluorescent Guided Robotic Surgery for Cancer of the Gastroesophageal Junction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, JENS OSTERKAMP, PhD fellow, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-19041735
Record Dates: First submitted 2019-08-01; First posted 2019-09-27 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Stomach Neoplasms; Surgery
Keywords: Gastric Conduit; Cardia resection; Indocyanine Green; quantative perfusion
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grupp 1 (Active Comparator): Patients will be allocated to preserving the right gastric artery during the resection of GEJ cancer.
  Interventions: Diagnostic Test: Indocyanine Green
- Grupp 2 (Active Comparator): Patients will be allocated to an extensive lymphatic resection (ligating the right gastric artery) during the resection of GEJ cancer.
  Interventions: Diagnostic Test: Indocyanine Green

INTERVENTIONS:
Diagnostic Test: Indocyanine Green — Using Q-ICG perfusion of the remaining Gastric Conduit will be compared

SUMMARY:
The investigators also aim to use our previously described quantifying method (q-ICG), to evaluate changes in gastric perfusion, during resection of cancer in the gastroesophageal junction (GEJ) and if a change in the operative technique influences microvascular flow in the gastroesophageal (GE) anastomosis.

DETAILED DESCRIPTION:
2. Introduction

2.1 Adenocarcinoma of the gastroesophageal tract Adenocarcinoma of the gastroesophageal tract, including the esophagus, stomach, and gastroesophageal junction (GEJ) is a growing clinical challenge worldwide due to the increasing incidence and poor prognosis. Current management of resectable GEJ cancer involves comprehensive diagnostic procedures followed by standardized treatment with surgery and pre- and postoperative chemotherapy.

At our department, 90 patients are annually treated for resectable cancer of the GEJ. The surgery comprises of an Ivor Lewis procedure with either open or robot-assisted mobilization of the stomach with limited (D1+) lymphadenectomy and creation of the gastric conduit and pyloroplasty (2). Here, the creation of the gastric conduit involves partial preservation of the right gastric artery. The right gastric artery is ligated approximately half way up the lesser curvature, and the remaining conduit stapled (figure 1). Theoretically, the preservation of both the gastro-epiploic and right gastric artery should result in improved vascular patency and blood supply to the anastomosis. The theoretical advantages of preserving the right gastric artery may have some oncological drawbacks as placing the line of resection half way up the lesser curvature allows for a limited lymph node (LN) dissection, leaving behind some tissue comprising of LN station number 3b and 5 (figure 1). Lymph node metastasis is a significant prognostic factor in gastroesophageal cancer, and the American Joint Committee on Cancer recommends an extensive lymphadenectomy to achieve accurate N staging.

In contrast, the creation of a gastric tube by serial applications of a linear-cutting stapling device parallel to the greater curvature (ligating the right gastric artery) could generate a larger LN harvest, but this could be at the expense of anastomotic and conduit perfusion. A retrospective series noted an increase in gastric tip necrosis and neck leaks with intrathoracic extension when a narrower gastric tube (3 to 4 cm) was used. Contrary, several randomized trials, and cohort studies have been conducted regarding the size of the gastric tube with no differences in anastomotic leakage rates being reported. However, the consensus is that a gastric tube of five cm width in both open and minimal invasive oesophagostomy is the optimal size. No difference in the rates of anastomotic leakage, anastomotic stenosis, or delayed gastric emptying has been seen between ligating or preserving the right gastric artery. Thus, both ligating and preserving the right gastric artery are considered viable surgical options.

Figure 1. A) Schematic image of the gastric blood vessels. B) Resection when ligating the right gastric artery, C) Resektion when preserving the right gastric artery. D) Schematic image and partial lymphatic overview, circled are lymph node stations 3b. and 5. resected in "B" and left behind in "C".

2.2 Fluorescence guided surgery with Indocyanine Green. Fluorescence guided surgery enables visualization of structures that are otherwise hidden from the naked human eye. A fluorescent contrast agent is used, often Indocyanine Green (ICG), and by illuminating the tissue with near-infrared light, the excited ICG can be detected by a camera with an optical filter. ICG is a tricarbocyanine dye with extremely few adverse events, a short half-life, it is metabolized exclusively in the liver, and excreted unchanged in the bile. The safety of ICG is well established, and it is used routinely in surgical clinics worldwide and has also in recent years gained popularity with regards to oncological surgery.

ICG binds to plasma proteins after intravenous injection, and by illuminating the tissue with near-infrared red light the fluorescence signal over time during first passage past tissue is considered proportional to microvascular flow, i.e., perfusion. Assessing gastrointestinal blood supply is a challenging task, even for experienced surgeons. Of specific concern is the vascular supply of the anastomosis since poor blood supply is a significant risk factor for anastomotic leakage. An esophagectomy is associated with an anastomotic leak rate of approximately 5 to 25 %. Anastomotic leakage after esophagectomy is a severe complication and associated with up to 17 % 30-day mortality. As ICG angiography allows for real-time visualization of visceral perfusion, an inadequate vascularisation of the anastomosis (despite satisfactory macroscopic appearance) can be detected and addressed intraoperatively. Thus, the use of perioperative ICG angiography has been shown to lower the risk of anastomotic leakage.

A study from our group evaluated intraoperative changes in the gastric microcirculation with laser speckle contrast imaging (LSCI) during Ivor-Lewis esophagectomy. A decreased microcirculation at the gastric corpus by 25% during mobilization of the stomach to the thorax was found. Also, ICG fluorescent intensity, as a sign of reduced perfusion, has been shown to drop after the formation of the gastric conduit and yet again before anastomosis formation compared with baseline values. This decrease was not detectable macroscopically in normal white light. However, macroscopic ICG assessments are useful as the speed of blood flow along the gastric conduit wall (visually assessed with ICG) could help predict the risk of anastomotic leakage after esophagectomy. Still, cut-off values for quantitative anastomotic perfusion associated with anastomotic leakage after resection of GEJ cancer is lacking. In conclusion, assuring adequate conduit perfusion is mandatory, and ICG angiography has been proven to be a viable aid in this regard.

Indocyanine Green retention in LNs has been shown to predict malignant content. In patients with esophageal- and GEJ cancer, a submucosal endoscopic ICG injection allowed the visualization of the tumor's lymphatic drainage. This visualization, could advance the diagnostics of malignant spread, increase lymph node harvest, and significantly affecting the choice of surgical resection.

The investigators have developed an ICG quantification algorithm which has been validated and described earlier. This algorithm has now been incorporated into a touch screen tablet, allowing for live perioperative quantitative perfusion assessments with ICG (q-ICG). A color-coded map of perfusion intensity is provided as an overlay on the white light visualized tissue (Figure 2). Previously, the quantification measurements had to be performed via analyses of video-recordings after the procedure. The investigators believe that q-ICG has the potential to improve intraoperative evaluation of tissue viability further and as such, improve the surgical plan and outcome in patients with GEJ cancer. In a feasibility study of ten patients undergoing GEJ-resection, significant alterations of optimal perfusion points selected by surgeons were found when comparing points selected in white light, ICG, and q-ICG.

In this trial, intravenous ICG injections will be used to evaluate conduit, and anastomotic perfusion and peritumoral intramucosal ICG injections will be used to evaluate a potential improvement in LN detection and harvest. Lymph node quantitative fluorescents will be compared with histological findings.

Figure 2. Gastric conduit after pull-up to the thorax viewed by white light, Near-Infrared Light (ICG) and with q-ICG overlay.

2.3 Aim The investigators aim to compare quantitative gastric conduit and anastomotic perfusion when preserving or ligating the right gastric artery. Further, the investigators wish to investigate weather peritumoral ICG injection will allow for additional lymph node visualization and harvest and examine the correlation between quantitative ICG fluorescents and histological findings.

2.4 Hypothesis The investigators hypothesize that ligating the right gastric artery will result in lesser perfusion of the gastric conduit and anastomosis. Further, the investigators hypothesize that peritumoral ICG injection will improve the identification of regional lymph nodes and potentially improve staging and the extent of lymphadenectomy.

3. Methods 3.1 Study design A randomized clinical trial comparing the effect of two different robotic-assisted surgical techniques for gastric conduit construction on conduit and anastomotic perfusion in patients with GEJ cancer. Patients will be allocated either to preserving the right gastric artery or to an extensive lymphatic resection (ligating the right gastric artery). Before and after the creation of the gastric conduit, and after the creation of the GE anastomosis, perfusion will be assessed with q-ICG.

The sample size calculation is based on estimating prediction models describing the relationship between the vascular ligation and gastric perfusion using linear regression. The investigators expect a reduced perfusion by 17%. The desired sample size is therefore n=70 (35 + 35), (effect 10%, SD 15%, Power 80%, alpha 0.05). Prospective evaluations of the surgical outcome will be recorded, by means of anastomotic leakage rates (verified endoscopically or radiologically), delayed gastric emptying (verified with barium swallow examination and/or endoscopy), and other postoperative complications including mortality. Also, the relationship between the quantified fluorescence of LNs and the pathology result will be examined in vivo and in vitro. The trial will be conducted in accordance with the CONSORT guidelines.

3.4 Recruitment Patients will be approached in the out-patient clinic. They will be informed orally, and written information will be provided. Written informed consent will be obtained from all patients before the procedure. All patients are informed of the possibility of withdrawal of their consent at any time during the trial without any consequence for the operation of their treatment. First, after written consent will inclusion in the study be possible.

3.5 Randomization The investigators wish to include 70 patients; 70 envelopes will be prepared each containing a "ligation" (n=35) or "preservation" (n=35) note. These seventy envelopes will be prepared and sealed by the trial investigator. A trial assistant will then mark these envelopes 1-70 at random using a number generator. Once the surgical set up is in place, one envelope will be chosen for each patient using a number generator, and the group allocation will be acquired. This patient CRP and Trial number will be saved on a secure server (L:drev). Separately the trial number and clinically relevant data will be stored on a secure server (V:drev).

3.6 Indocyanine green Indocyanine green is a well-described nontoxic tricarbocyanine dye used for decades in ophthalmology, cardiology, and hepatology. Very few mild adverse reactions have been reported, but caution in patients with thyrotoxicosis, allergy towards iodine or indocyanine green should be made. When injected, it binds to blood lipoproteins and is solely metabolized by the liver and excreted in the bile, with a short half-life of approximately 4-5 minutes. Indocyanine green is already used as a routine in many specialties; here among surgery, ophthalmology, hepatology, and cardiology.

3.7 Surgical procedure and perfusion assessment

3.7.1 Resection of the gastroesophageal junction The patient is placed under general anesthesia and, using a standard adult endoscope, 2 mL of ICG doubly diluted in sterile water (5 mg/mL) is injected into the submucosa at the four quadrants around the tumor (0.5 mL for each injection). The robotic setup is after that completed. Based on previous studies, the time from injection to lymph node visualization is approximated to 10-30 min.

After the initial presentation of the stomach is acquired, a bolus of ICG (0.2 mg/kg body weight) will be injected intravenously and flushed with 5 mL of saline. The ROIs will then be assessed with q-ICG. The anesthetic protocol will to this point match that of the setting during the screening laparoscopy. The q-ICG assessments then repeated after the dissection, division of the feeding blood vessels and the creation of the conduit. Finally, once the gastroesophageal anastomosis is completed a q-ICG assessment of anastomotic perfusion will be performed.

3.7.2 Fluorescence angiography The GEJ resection will be carried out with the da Vinci® robot, (Intuitive Surgical Systems, Sunnyvale, CA, USA) and the fluorescent angiography will be performed using the infrared endoscopic equipment on the da Vinci® robotic system (Firefly® in the DaVinci Xi).

3.8 Statistics Comparison of the gastric and anastomotic perfusion between groups will be performed using the Mann Whitney U test or a paired sample t-test depending on either a non- or parametric nature of the data. Between-group differences in continuous variables were assessed using analysis of variance, while those in categorical variable were assessed using pooled relative risk with 95% confidence interval (CI). A P-value < 0.05 will be considered significant. Statistic evaluation will be performed using IBM SPSS Statistics © (v 22.0 SPSS Inc. Chicago, IL, USA).

4. Adverse events, risks, and disadvantages Adverse events associated with the use of ICG are rare, and severe anaphylactic reactions are extremely rare. However, safety precautions will be made by excluding patients with allergy to iodine, ICG, or shellfish. Also, the investigators will not include patients with severe kidney and liver insufficiency, thyrotoxicosis, and pregnant or lactating women. The total dose of dye injected will be kept well below the recommended 2 mg/kg. There are no data available describing the signs, symptoms, or laboratory findings accompanying overdosage. The LD50 after I.V. administration ranges between 60 and 80 mg/kg in mice, 50 and 70 mg/kg in rats and 50 and 80 mg/kg in rabbits.

No difference in the rates of anastomotic leakage, anastomotic stenosis, or delayed gastric emptying has been seen between ligating or preserving the right gastric artery, and both are considered viable surgical options.

5. Patient data Upon meeting in the out-patient clinic, the patients will be informed about an ongoing study and asked if they wish further information. If accepted the principle investigator will be called and to briefly inform the patient about the project, and ask about allergy towards; iodine, indocyanine green or shellfish, liver insufficiency, thyrotoxicosis, pregnancy or lactation. If no allergies exist, the patient will then receive written, and oral information about the project and a follow-up telephone call regarding inclusion will be held. If interested in participation, the patient will supply the principle investigator with written consent. The written consent provides with access to obtain information in the patient's electronic journal. This, to see information about the subject's health and the course during hospitalization, necessary as part of the research project. Including self-control, quality control, and monitoring, which are obligatory. Data obtained from electronic patient records are registered prospectively and pseudo-anonymized in a database and kept at the secure server provided by Region Hovedstaden (V:drev). Thus, data in this database may not be identified back to the patient without access to a patient participation list linking patient identification number and the pseudo anonymization number. This participation list will be stored in another folder on the secure server provided by the Region Hovedstaden (L:drev). Only the principle investigator, supervisors and will have access to these folders and files. The law on the processing of personal data (Persondataloven) will, of course, be followed. No data will be sent to other countries. Permission from the national data protection (Datatilsynet) agency will be obtained.

6. Ethical considerations Approval from the regional ethical committee and the national data protection agency will be in place before initiating the study.

ICG is a safe and non-toxic fluorescent dye as described and has been used for decades in ophthalmology, cardiology, and hepatology. Very few adverse reactions are reported. Patients may withdraw from the study at any time. The patients participating in the study will not be paid to participate. Both preserving and ligation the right gastric artery are considered safe and viable surgical approaches.

7. Publication The investigators aim to publish negative, positive, and inconclusive results in international reputed surgical journals, possibly as open access with Jens Osterkamp as the primary author. Also, the investigators will present the work at national and/or international surgical conferences and meetings to share the findings with a large crowd of clinicians and researchers.

8. Timeframe The study will be initiated as soon as the investigators have approval from the ethical committee and the national data protection agency. Hopefully, starting in early 2020, and completed ultimo 2023.

9. Economy This study is a part of the principle investigators Ph.-thesis. Salary and experimental cost will be cover by a grant provided by Medtronic. With regards to study design, realization, and presentation, the research group has complete autonomy. No remuneration will be given to patients participating in the trial. The principal investigator has in collaboration with the project group initiated the project. There are no financial interests for the project group in this project. Equipment (tablet, video-capture device, laparoscopic equipment, surgical robot) is already present in the department. If additional support is granted, the name of the foundation(s), size of the amount, any relation between the grant provider and investigators, as well as any requirements of the grants will be announced to the committee and project participants (patients).

10. Insurance Patients will be covered by the national Danish patient insurance.

ELIGIBILITY:
Inclusion Criteria:

* Patients (above 18 years) scheduled for planned open or robot-assisted resection of gastroesophageal junction cancer.

Exclusion Criteria:

* Allergy towards; iodine, indocyanine green or shellfish
* Severe liver insufficiency
* Thyrotoxicosis
* Nephropathy requiring dialysis
* Pregnancy or lactation
* Legally incompetent for any reason
* Withdrawal of inclusion consent at any time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2021-10-13 (Actual)

PRIMARY OUTCOMES:
perfusion assessment | The perfussion assesment takes 3-5min.
  The primary endpoint is the difference in conduit- and anastomotic perfusion between the two groups. The perfusion will be measured intraoperativly using q-ICG.

SECONDARY OUTCOMES:
Lymph node resektion | Caculated after the return of pathology report. The patients will be followed 30 days after surgery
  Number of lymph nodes harvested
short term surgical outcome | Patients will be follow for 30 days after surgery
  Clavien- Dindo Index
short term surgical outcome | Patients will be follow for 30 days after surgery
  Comprehensive Complication Index
short term surgical outcome | Patients will be follow for 30 days after surgery
  length of hospital stay, in days.
short term surgical outcome | Patients will be follow for 30 days after surgery
  Complications will be defined as any deviation from the normal postoperative course. This definition also takes into account asymptomatic complications such as arrhythmia, ECG.
short term surgical outcome | Patients will be follow for 30 days after surgery
  Complications will be defined as any deviation from the normal postoperative course. This definition also takes into account asymptomatic complications such as and atelectasis, chest x ray
short term surgical outcome | Patients will be follow for 30 days after surgery
  Complications will be defined as any deviation from the normal postoperative course. This definition also takes into account asymptomatic complications such affected blood test.
Anastomotic leakage | the patients will be follow 30 days after surgery
  Cut-off values for q-ICG anastomotic perfusion associated with anastomotic leakage. Diagnosed on x-ray or clinical examination.

CONTACTS AND LOCATIONS:
Overall Officials: Jens TF Osterkamp, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chiappa A, Andreoni B, Dionigi R, Spaggiari L, Foschi D, Polvani G, Orecchia R, Fazio N, Pravettoni G, Cossu ML, Galetta D, Venturino M, Ferrari C, Macone L, Crosta C, Bonanni B, Biffi R. A rationale multidisciplinary approach for treatment of esophageal and gastroesophageal junction cancer: Accurate review of management and perspectives. Crit Rev Oncol Hematol. 2018 Dec;132:161-168. doi: 10.1016/j.critrevonc.2018.10.002. Epub 2018 Oct 13. PMID 30447922
- [Background] Kofoed SC, Calatayud D, Jensen LS, Helgstrand F, Achiam MP, De Heer P, Svendsen LB; Danish Esophageal, Cardia and Stomach Cancer Group. Intrathoracic anastomotic leakage after gastroesophageal cancer resection is associated with increased risk of recurrence. J Thorac Cardiovasc Surg. 2015 Jul;150(1):42-8. doi: 10.1016/j.jtcvs.2015.04.030. Epub 2015 Apr 21. PMID 25986493
- [Background] Akiyama H, Miyazono H, Tsurumaru M, Hashimoto C, Kawamura T. Use of the stomach as an esophageal substitute. Ann Surg. 1978 Nov;188(5):606-10. doi: 10.1097/00000658-197811000-00004. PMID 718285
- [Background] Ndoye JM, Dia A, Ndiaye A, Fall B, Diop M, Ndiaye A, Sow ML. Arteriography of three models of gastric oesophagoplasty: the whole stomach, a wide gastric tube and a narrow gastric tube. Surg Radiol Anat. 2006 Oct;28(5):429-37. doi: 10.1007/s00276-006-0129-5. Epub 2006 Jul 19. PMID 16850349
- [Background] Collard JM, Tinton N, Malaise J, Romagnoli R, Otte JB, Kestens PJ. Esophageal replacement: gastric tube or whole stomach? Ann Thorac Surg. 1995 Aug;60(2):261-6; discussion 267. doi: 10.1016/0003-4975(95)00411-d. PMID 7646084
- [Background] Nussbaum DP, Pappas TN, Perez A. Laparoscopic Total Gastrectomy in the Western Patient Population: Tips, Techniques, and Evidence-based Practice. Surg Laparosc Endosc Percutan Tech. 2015 Dec;25(6):455-61. doi: 10.1097/SLE.0000000000000210. PMID 26492457
- [Background] Egner, J. R. AJCC Cancer Staging Manual. JAMA 304, 1726 (2010
- [Background] Boyle NH, Pearce A, Hunter D, Owen WJ, Mason RC. Intraoperative scanning laser Doppler flowmetry in the assessment of gastric tube perfusion during esophageal resection. J Am Coll Surg. 1999 May;188(5):498-502. doi: 10.1016/s1072-7515(99)00016-2. PMID 10235577
- [Background] Luketich JD, Alvelo-Rivera M, Buenaventura PO, Christie NA, McCaughan JS, Litle VR, Schauer PR, Close JM, Fernando HC. Minimally invasive esophagectomy: outcomes in 222 patients. Ann Surg. 2003 Oct;238(4):486-94; discussion 494-5. doi: 10.1097/01.sla.0000089858.40725.68. PMID 14530720
- [Background] Shu YS, Sun C, Shi WP, Shi HC, Lu SC, Wang K. Tubular stomach or whole stomach for esophagectomy through cervico-thoraco-abdominal approach: a comparative clinical study on anastomotic leakage. Ir J Med Sci. 2013 Sep;182(3):477-80. doi: 10.1007/s11845-013-0917-y. Epub 2013 Feb 10. PMID 23397501
- [Background] Bemelman WA, Taat CW, Slors JF, van Lanschot JJ, Obertop H. Delayed postoperative emptying after esophageal resection is dependent on the size of the gastric substitute. J Am Coll Surg. 1995 Apr;180(4):461-4. PMID 7719551
- [Background] Tabira Y, Sakaguchi T, Kuhara H, Teshima K, Tanaka M, Kawasuji M. The width of a gastric tube has no impact on outcome after esophagectomy. Am J Surg. 2004 Mar;187(3):417-21. doi: 10.1016/j.amjsurg.2003.12.008. PMID 15006575
- [Background] Zhang C, Wu QC, Hou PY, Zhang M, Li Q, Jiang YJ, Chen D. Impact of the method of reconstruction after oncologic oesophagectomy on quality of life--a prospective, randomised study. Eur J Cardiothorac Surg. 2011 Jan;39(1):109-14. doi: 10.1016/j.ejcts.2010.04.032. Epub 2010 Jun 9. PMID 20538475
- [Background] Collard JM, Romagnoli R, Otte JB, Kestens PJ. The denervated stomach as an esophageal substitute is a contractile organ. Ann Surg. 1998 Jan;227(1):33-9. doi: 10.1097/00000658-199801000-00005. PMID 9445107
- [Background] Pennathur A, Awais O, Luketich JD. Technique of minimally invasive Ivor Lewis esophagectomy. Ann Thorac Surg. 2010 Jun;89(6):S2159-62. doi: 10.1016/j.athoracsur.2010.03.069. PMID 20494002
- [Background] Zhang W, Yu D, Peng J, Xu J, Wei Y. Gastric-tube versus whole-stomach esophagectomy for esophageal cancer: A systematic review and meta-analysis. PLoS One. 2017 Mar 7;12(3):e0173416. doi: 10.1371/journal.pone.0173416. eCollection 2017. PMID 28267808
- [Background] Hartwig W, Strobel O, Schneider L, Hackert T, Hesse C, Buchler MW, Werner J. Fundus rotation gastroplasty vs. Kirschner-Akiyama gastric tube in esophageal resection: comparison of perioperative and long-term results. World J Surg. 2008 Aug;32(8):1695-702. doi: 10.1007/s00268-008-9648-z. PMID 18553046
- [Background] Garski TR, Staller BJ, Hepner G, Banka VS, Finney RA Jr. Adverse reactions after administration of indocyanine green. JAMA. 1978 Aug 18;240(7):635. doi: 10.1001/jama.240.7.635b. No abstract available. PMID 671679
- [Background] Alander JT, Kaartinen I, Laakso A, Patila T, Spillmann T, Tuchin VV, Venermo M, Valisuo P. A review of indocyanine green fluorescent imaging in surgery. Int J Biomed Imaging. 2012;2012:940585. doi: 10.1155/2012/940585. Epub 2012 Apr 22. PMID 22577366
- [Background] Baiocchi GL, Diana M, Boni L. Indocyanine green-based fluorescence imaging in visceral and hepatobiliary and pancreatic surgery: State of the art and future directions. World J Gastroenterol. 2018 Jul 21;24(27):2921-2930. doi: 10.3748/wjg.v24.i27.2921. PMID 30038461
- [Background] Pommergaard HC, Achiam MP, Burcharth J, Rosenberg J. Impaired blood supply in the colonic anastomosis in mice compromises healing. Int Surg. 2015 Jan;100(1):70-6. doi: 10.9738/INTSURG-D-13-00191.1. PMID 25594642
- [Background] Kruschewski M, Rieger H, Pohlen U, Hotz HG, Buhr HJ. Risk factors for clinical anastomotic leakage and postoperative mortality in elective surgery for rectal cancer. Int J Colorectal Dis. 2007 Aug;22(8):919-27. doi: 10.1007/s00384-006-0260-0. Epub 2007 Jan 27. PMID 17260142
- [Background] Kim MJ, Shin R, Oh HK, Park JW, Jeong SY, Park JG. The impact of heavy smoking on anastomotic leakage and stricture after low anterior resection in rectal cancer patients. World J Surg. 2011 Dec;35(12):2806-10. doi: 10.1007/s00268-011-1286-1. PMID 21959931
- [Background] Fawcett A, Shembekar M, Church JS, Vashisht R, Springall RG, Nott DM. Smoking, hypertension, and colonic anastomotic healing; a combined clinical and histopathological study. Gut. 1996 May;38(5):714-8. doi: 10.1136/gut.38.5.714. PMID 8707117
- [Background] Kassis ES, Kosinski AS, Ross P Jr, Koppes KE, Donahue JM, Daniel VC. Predictors of anastomotic leak after esophagectomy: an analysis of the society of thoracic surgeons general thoracic database. Ann Thorac Surg. 2013 Dec;96(6):1919-26. doi: 10.1016/j.athoracsur.2013.07.119. Epub 2013 Sep 24. PMID 24075499
- [Background] Alanezi K, Urschel JD. Mortality secondary to esophageal anastomotic leak. Ann Thorac Cardiovasc Surg. 2004 Apr;10(2):71-5. PMID 15209546
- [Background] Udagawa H, Akiyama H. Surgical treatment of esophageal cancer: Tokyo experience of the three-field technique. Dis Esophagus. 2001;14(2):110-4. doi: 10.1046/j.1442-2050.2001.00166.x. PMID 11553219
- [Background] Ando N, Ozawa S, Kitagawa Y, Shinozawa Y, Kitajima M. Improvement in the results of surgical treatment of advanced squamous esophageal carcinoma during 15 consecutive years. Ann Surg. 2000 Aug;232(2):225-32. doi: 10.1097/00000658-200008000-00013. PMID 10903602
- [Background] Ryan CE, Paniccia A, Meguid RA, McCarter MD. Transthoracic Anastomotic Leak After Esophagectomy: Current Trends. Ann Surg Oncol. 2017 Jan;24(1):281-290. doi: 10.1245/s10434-016-5417-7. Epub 2016 Jul 12. PMID 27406098
- [Background] Chadi SA, Fingerhut A, Berho M, DeMeester SR, Fleshman JW, Hyman NH, Margolin DA, Martz JE, McLemore EC, Molena D, Newman MI, Rafferty JF, Safar B, Senagore AJ, Zmora O, Wexner SD. Emerging Trends in the Etiology, Prevention, and Treatment of Gastrointestinal Anastomotic Leakage. J Gastrointest Surg. 2016 Dec;20(12):2035-2051. doi: 10.1007/s11605-016-3255-3. Epub 2016 Sep 16. PMID 27638764
- [Background] Mangano A, Fernandes E, Gheza F, Bustos R, Chen LL, Masrur M, Giulianotti PC. Near-Infrared Indocyanine Green-Enhanced Fluorescence and Evaluation of the Bowel Microperfusion During Robotic Colorectal Surgery: a Retrospective Original Paper. Surg Technol Int. 2019 May 15;34:93-100. PMID 30716160
- [Background] Zehetner J, DeMeester SR, Alicuben ET, Oh DS, Lipham JC, Hagen JA, DeMeester TR. Intraoperative Assessment of Perfusion of the Gastric Graft and Correlation With Anastomotic Leaks After Esophagectomy. Ann Surg. 2015 Jul;262(1):74-8. doi: 10.1097/SLA.0000000000000811. PMID 25029436
- [Background] Mangano A, Gheza F, Chen LL, Minerva EM, Giulianotti PC. Indocyanine Green (Icg)-Enhanced Fluorescence for Intraoperative Assessment of Bowel Microperfusion During Laparoscopic and Robotic Colorectal Surgery: The Quest for Evidence-Based Results. Surg Technol Int. 2018 Jun 1;32:101-104. PMID 29611153
- [Background] Gossedge G, Vallance A, Jayne D. Diverse applications for near infra-red intraoperative imaging. Colorectal Dis. 2015 Oct;17 Suppl 3:7-11. doi: 10.1111/codi.13023. PMID 26394736
- [Background] Watanabe J, Ishibe A, Suwa Y, Suwa H, Ota M, Kunisaki C, Endo I. Indocyanine green fluorescence imaging to reduce the risk of anastomotic leakage in laparoscopic low anterior resection for rectal cancer: a propensity score-matched cohort study. Surg Endosc. 2020 Jan;34(1):202-208. doi: 10.1007/s00464-019-06751-9. Epub 2019 Mar 14. PMID 30877565
- [Background] Sujatha-Bhaskar S, Jafari MD, Stamos MJ. The Role of Fluorescent Angiography in Anastomotic Leaks. Surg Technol Int. 2017 Jul 25;30:83-88. PMID 28277591
- [Background] Ambrus R, Svendsen LB, Secher NH, Runitz K, Frederiksen HJ, Svendsen MB, Siemsen M, Kofoed SC, Achiam MP. A reduced gastric corpus microvascular blood flow during Ivor-Lewis esophagectomy detected by laser speckle contrast imaging technique. Scand J Gastroenterol. 2017 Apr;52(4):455-461. doi: 10.1080/00365521.2016.1265664. Epub 2016 Dec 15. PMID 27973925
- [Background] Ishige F, Nabeya Y, Hoshino I, Takayama W, Chiba S, Arimitsu H, Iwatate Y, Yanagibashi H. Quantitative Assessment of the Blood Perfusion of the Gastric Conduit by Indocyanine Green Imaging. J Surg Res. 2019 Feb;234:303-310. doi: 10.1016/j.jss.2018.08.056. Epub 2018 Oct 23. PMID 30527489
- [Background] Koyanagi K, Ozawa S, Oguma J, Kazuno A, Yamazaki Y, Ninomiya Y, Ochiai H, Tachimori Y. Blood flow speed of the gastric conduit assessed by indocyanine green fluorescence: New predictive evaluation of anastomotic leakage after esophagectomy. Medicine (Baltimore). 2016 Jul;95(30):e4386. doi: 10.1097/MD.0000000000004386. PMID 27472732
- [Background] Jansen SM, de Bruin DM, van Berge Henegouwen MI, Strackee SD, Veelo DP, van Leeuwen TG, Gisbertz SS. Optical techniques for perfusion monitoring of the gastric tube after esophagectomy: a review of technologies and thresholds. Dis Esophagus. 2018 Jun 1;31(6). doi: 10.1093/dote/dox161. PMID 29701760
- [Background] Pop CF, Veys I, Gomez Galdon M, Moreau M, Larsimont D, Donckier V, Bourgeois P, Liberale G. Ex vivo indocyanine green fluorescence imaging for the detection of lymph node involvement in advanced-stage ovarian cancer. J Surg Oncol. 2018 Dec;118(7):1163-1169. doi: 10.1002/jso.25263. Epub 2018 Oct 7. PMID 30293250
- [Background] Liberale G, Vankerckhove S, Caldon MG, Ahmed B, Moreau M, Nakadi IE, Larsimont D, Donckier V, Bourgeois P; Group R&D for the Clinical Application of Fluorescence Imaging of the Jules Bordet's Institute.. Fluorescence Imaging After Indocyanine Green Injection for Detection of Peritoneal Metastases in Patients Undergoing Cytoreductive Surgery for Peritoneal Carcinomatosis From Colorectal Cancer: A Pilot Study. Ann Surg. 2016 Dec;264(6):1110-1115. doi: 10.1097/SLA.0000000000001618. PMID 27828822
- [Background] Digonnet A, van Kerckhove S, Moreau M, Willemse E, Quiriny M, Ahmed B, de Saint Aubain N, Andry G, Bourgeois P. Near infrared fluorescent imaging after intravenous injection of indocyanine green during neck dissection in patients with head and neck cancer: A feasibility study. Head Neck. 2016 Apr;38 Suppl 1:E1833-7. doi: 10.1002/hed.24331. Epub 2015 Dec 24. PMID 26699164
- [Background] Xia L, Zeh R, Mizelle J, Newton A, Predina J, Nie S, Singhal S, Guzzo TJ. Near-infrared Intraoperative Molecular Imaging Can Identify Metastatic Lymph Nodes in Prostate Cancer. Urology. 2017 Aug;106:133-138. doi: 10.1016/j.urology.2017.04.020. Epub 2017 Apr 21. PMID 28438626
- [Background] Satou S, Ishizawa T, Masuda K, Kaneko J, Aoki T, Sakamoto Y, Hasegawa K, Sugawara Y, Kokudo N. Indocyanine green fluorescent imaging for detecting extrahepatic metastasis of hepatocellular carcinoma. J Gastroenterol. 2013 Oct;48(10):1136-43. doi: 10.1007/s00535-012-0709-6. Epub 2012 Nov 20. PMID 23179608
- [Background] Schlottmann F, Barbetta A, Mungo B, Lidor AO, Molena D. Identification of the Lymphatic Drainage Pattern of Esophageal Cancer with Near-Infrared Fluorescent Imaging. J Laparoendosc Adv Surg Tech A. 2017 Mar;27(3):268-271. doi: 10.1089/lap.2016.0523. Epub 2016 Dec 19. PMID 27992300
- [Background] Hachey KJ, Gilmore DM, Armstrong KW, Harris SE, Hornick JL, Colson YL, Wee JO. Safety and feasibility of near-infrared image-guided lymphatic mapping of regional lymph nodes in esophageal cancer. J Thorac Cardiovasc Surg. 2016 Aug;152(2):546-54. doi: 10.1016/j.jtcvs.2016.04.025. Epub 2016 Apr 11. PMID 27179838
- [Background] Nerup N, Andersen HS, Ambrus R, Strandby RB, Svendsen MBS, Madsen MH, Svendsen LB, Achiam MP. Quantification of fluorescence angiography in a porcine model. Langenbecks Arch Surg. 2017 Jun;402(4):655-662. doi: 10.1007/s00423-016-1531-z. Epub 2016 Nov 15. PMID 27848028
- [Background] Simonsen C, de Heer P, Bjerre ED, Suetta C, Hojman P, Pedersen BK, Svendsen LB, Christensen JF. Sarcopenia and Postoperative Complication Risk in Gastrointestinal Surgical Oncology: A Meta-analysis. Ann Surg. 2018 Jul;268(1):58-69. doi: 10.1097/SLA.0000000000002679. PMID 29373365
- [Background] Horowitz M, Neeman E, Sharon E, Ben-Eliyahu S. Exploiting the critical perioperative period to improve long-term cancer outcomes. Nat Rev Clin Oncol. 2015 Apr;12(4):213-26. doi: 10.1038/nrclinonc.2014.224. Epub 2015 Jan 20. PMID 25601442
- [Background] Trencheva K, Morrissey KP, Wells M, Mancuso CA, Lee SW, Sonoda T, Michelassi F, Charlson ME, Milsom JW. Identifying important predictors for anastomotic leak after colon and rectal resection: prospective study on 616 patients. Ann Surg. 2013 Jan;257(1):108-13. doi: 10.1097/SLA.0b013e318262a6cd. PMID 22968068
- [Background] Thompson SK, Chang EY, Jobe BA. Clinical review: Healing in gastrointestinal anastomoses, part I. Microsurgery. 2006;26(3):131-6. doi: 10.1002/micr.20197. PMID 16518804
- [Background] Otto JM, Plumb JOM, Wakeham D, Clissold E, Loughney L, Schmidt W, Montgomery HE, Grocott MPW, Richards T. Total haemoglobin mass, but not haemoglobin concentration, is associated with preoperative cardiopulmonary exercise testing-derived oxygen-consumption variables. Br J Anaesth. 2017 May 1;118(5):747-754. doi: 10.1093/bja/aew445. PMID 28510737
- [Background] Lundby C, Montero D, Joyner M. Biology of VO2 max: looking under the physiology lamp. Acta Physiol (Oxf). 2017 Jun;220(2):218-228. doi: 10.1111/apha.12827. Epub 2016 Nov 25. PMID 27888580
- [Background] Christensen JF, Jones LW, Tolver A, Jorgensen LW, Andersen JL, Adamsen L, Hojman P, Nielsen RH, Rorth M, Daugaard G. Safety and efficacy of resistance training in germ cell cancer patients undergoing chemotherapy: a randomized controlled trial. Br J Cancer. 2014 Jul 8;111(1):8-16. doi: 10.1038/bjc.2014.273. Epub 2014 May 27. PMID 24867693
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c869. doi: 10.1136/bmj.c869. No abstract available. PMID 20332511
- [Background] Owens SL. Indocyanine green angiography. Br J Ophthalmol. 1996 Mar;80(3):263-6. doi: 10.1136/bjo.80.3.263. No abstract available. PMID 8703866
- [Background] Spinoglio G, Bertani E, Borin S, Piccioli A, Petz W. Green indocyanine fluorescence in robotic abdominal surgery. Updates Surg. 2018 Sep;70(3):375-379. doi: 10.1007/s13304-018-0585-6. Epub 2018 Aug 29. PMID 30159820
- [Background] Herrera-Almario G, Patane M, Sarkaria I, Strong VE. Initial report of near-infrared fluorescence imaging as an intraoperative adjunct for lymph node harvesting during robot-assisted laparoscopic gastrectomy. J Surg Oncol. 2016 Jun;113(7):768-70. doi: 10.1002/jso.24226. Epub 2016 Mar 29. PMID 27021142
- [Derived] Osterkamp J, Strandby R, Nerup N, Svendsen MB, Svendsen LB, Achiam M. Intraoperative near-infrared lymphography with indocyanine green may aid lymph node dissection during robot-assisted resection of gastroesophageal junction cancer. Surg Endosc. 2023 Mar;37(3):1985-1993. doi: 10.1007/s00464-022-09684-y. Epub 2022 Oct 21. PMID 36271062